CLINICAL TRIAL: NCT01522573
Title: Therapeutic Endoscopic Ultrasound (T-EUS) Guided Procedures in the Management of Gastrointestinal Disorders: A Multicenter Registry.
Brief Title: T-EUS for Gastrointestinal Disorders: A Multicenter Registry
Acronym: EUSERCPReg
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief, Advanced Endoscopy, Weill Medical College of Cornell University
Other Study IDs: 1111012016
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Cholangiocarcinoma; Pancreatic Cancer; Bile Duct Cancer; Biliary Stricture; Biliary Obstruction; Stent Obstruction; Proximal Duct Stricture; Distal Duct Stricture; Ampullary Cancer; Biliary Sphincter Stenosis; Impacted Stones; Chronic Pancreatitis; Peri-ampullary Diverticula; Altered Anatomy
Keywords: Cholangiocarcinoma; Pancreatic Cancer; Bile Duct Cancer; Biliary Stricture; Biliary obstruction; Stent obstruction; Proximal duct stricture; Distal duct stricture; Ampullary Cancer; Biliary sphincter stenosis; Impacted stones; Chronic pancreatitis; Peri-ampullary diverticula; Altered anatomy; Endoscopic ultrasound; Endoscopic Retrograde Cholangiopancreatography; Multicenter
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms; Bile Duct Neoplasms; Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EUS guided ERCP procedure group: Subjects who will undergo Endoscopic Ultrasound (EUS) guided Endoscopic retrograde cholangiopancreatography (ERCP) procedures for their pancreatico-biliary conditions.
  Interventions: Procedure: EUS guided ERCP

INTERVENTIONS:
Procedure: EUS guided ERCP — Endoscopic ultrasound guided (EUS) endoscopic retrograde cholangiopancreatography (ERCP)
  Other Names: EUS ERCP

SUMMARY:
The purpose of this registry is to record information and evaluate the impact of Endoscopic Ultrasound (EUS) Guided Endoscopic retrograde cholangiopancreatography (ERCP) on the management of pancreatico-biliary disorders. The registry will evaluate efficacy, safety and technical success of the Endoscopic Ultrasound (EUS)Guided Endoscopic retrograde cholangiopancreatography (ERCP) procedures. The safety and efficacy of various EUS-Guided ERCP procedures have been assessed in a series of studies.

This multi-center registry has been initiated:

* To document the impact of EUS-Guided ERCP procedures on the management of pancreatico-biliary disorders including malignancies.
* To assess the clinical and technical success rates of EUS-Guided ERCPs for diagnostic or therapeutic procedures.

Design is retrospective and prospective registry study.

Procedures that will be captured include:

1. EUS-Coils placement
2. EUS Glue injection
3. EUS-Fiducial placement
4. EUS-Neurolysis
5. EUS-Stent placement
6. EUS-alcohol injection
7. EUS-fluid collection, abscess or cavity drainage
8. EUS guided ductal drainage
9. EUS-guided Ablation
10. EUS-guided anastomosis 11. EUS Guided ERCP for gallbladder, pancreatic duct or biliary duct drainage

DETAILED DESCRIPTION:
Endoscopic Ultrasound (EUS) Guided Endoscopic retrograde cholangiopancreatography (ERCP) has become a therapeutic intervention for the management of biliary obstruction or pancreatic strictures related to chronic pancreatitis or other diseases. Successful biliary or pancreatic cannulation can be achieved in 90 to 97%. Failure to obtain biliary access can be related to operator experience, peri-ampullary diverticula, prior surgery (e.g., Billroth II anatomy), tumor involvement of the ampulla, biliary sphincter stenosis and impacted stones. In experienced hands, pancreatic duct cannulation fails in less than 10% of cases. This is primarily related to surgically altered anatomy or inflammation. Referral to a tertiary care center , percutaneous intrahepatic cholangiography (PTC) for biliary decompression , and surgical intervention are typically offered after a failed ERCP. Percutaneous intrahepatic cholangiography with subsequent percutaneous or endoscopic drainage has a morbidity of up to 32%. Surgery can also be associated with significant morbidity and mortality.

Endoscopic ultrasound (EUS) allows detailed imaging of the regional anatomy by approximating the frequency transducer to the region of interest. With the evolution of linear array and the ability to direct a needle within the field of interest, the therapeutic potential of EUS has reached new levels beyond fine needle aspiration (FNA), celiac plexus blocks and drainage of cystic lesions. The biliary and pancreatic systems, being in close proximity to the gastric or duodenal lumen, are a logical target for EUS in cases not accessible by ERCP. EUS-assisted cholangiopancreatography was described a decade ago. In order to validate these procedures and broaden its use beyond tertiary centers, it is crucial to understand its efficacy and success rate. The objective of the study is to evaluate retrospectively and prospectively the efficacy and safety of EUS-Guided ERCP procedures for the diagnosis and treatment of pancreatico-biliary disorders.

The purpose of this registry is to record information and evaluate the impact of EUS-Guided ERCP on the management of pancreatico-biliary disorders. The registry will evaluate efficacy, safety and technical success of the EUS-Guided ERCP procedures.

The involvement of multi-international sites is crucial- as the advanced endoscopists outside US are attempting similar complex EUS-Guided ERCPs for complicated pancreatico-biliary cases as their counterparts in US. However, because of the non-existence of a registry, these cases are often reported as isolated case series with remarkable technical similarities to case series in other countries.

The registry hopes to combine all such comparable cases and collect enough relevant data for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has undergone EUS-guided ERCP (Endoscopic Retrograde Cholangiopancreatography)for diagnosis or treatment of a pancreatico-biliary disorder.
* Above 18 years of age.

Exclusion Criteria:

* Any subject who has not undergone Endoscopic Ultrasound (EUS) guided Endoscopic retrograde cholangiopancreatography (ERCP).
* Below 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who has undergone Endoscopic Ultrasound (EUS) guided Endoscopic retrograde cholangiopancreatography (ERCP) procedure for diagnosis or treatment of a pancreatico-biliary disorder.
  Above 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-11; Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety | 3 years
  Documentation of Safety- Number of Participants with Adverse Events; Type, frequency and intensity of adverse events

SECONDARY OUTCOMES:
Efficacy | 3 years
  Documentation of efficacy: Technical and clinical success rates.
  * Technical Success rate will be derived from reported success or failure of technical feasibility and conduction of a specific EUS Guided ERCP procedure for a pancreatico-biliary condition.
  * Clinical success rate will be derived from reported of clinical success hallmarks such as biliary or pancreatic drainage, reduction in total bilirubin, formation of a fistula, immediate and eventual alleviation of symptoms or complaints within a specific period of time, etc. for that particular pancreatico-biliary disorder.
Survival duration | 3 years
  Documentation of response rates and overall survival duration.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- Weill Cornell Medical College, New York, New York, United States
- Prof. Dr. Everson L.A. Artifon, São Paulo, Brazil

REFERENCES:
- [Derived] Tyberg A, Kats D, Choi A, Gaidhane M, Nieto J, Kahaleh M. Endoscopic Ultrasound Guided Gastroenterostomy: What Is the Learning Curve? J Clin Gastroenterol. 2021 Sep 1;55(8):691-693. doi: 10.1097/MCG.0000000000001400. PMID 32740096
- [Derived] Kumta NA, Tyberg A, Bhagat VH, Siddiqui AA, Kowalski TE, Loren DE, Desai AP, Sarkisian AM, Brown EG, Karia K, Gaidhane M, Kedia P, Tarnasky PR, Patel U, Adler D, Taylor LJ, Petrone M, Arcidiacono P, Yachimski PS, Weine D, Sundararajan S, Deprez PH, Mouradides C, Ho S, Javed S, Easler JJ, Raijman I, Vazquez-Sequeiros E, Sawhney M, Berzin TM, Kahaleh M. EUS-guided drainage of pancreatic fluid collections using lumen apposing metal stents: An international, multicenter experience. Dig Liver Dis. 2019 Nov;51(11):1557-1561. doi: 10.1016/j.dld.2019.05.033. Epub 2019 Jul 2. PMID 31272934
- [Derived] Siddiqui A, Kunda R, Tyberg A, Arain MA, Noor A, Mumtaz T, Iqbal U, Loren DE, Kowalski TE, Adler DG, Saumoy M, Gaidhane M, Mallery S, Christiansen EM, Nieto J, Kahaleh M. Three-way comparative study of endoscopic ultrasound-guided transmural gallbladder drainage using lumen-apposing metal stents versus endoscopic transpapillary drainage versus percutaneous cholecystostomy for gallbladder drainage in high-risk surgical patients with acute cholecystitis: clinical outcomes and success in an International, Multicenter Study. Surg Endosc. 2019 Apr;33(4):1260-1270. doi: 10.1007/s00464-018-6406-7. Epub 2018 Sep 12. PMID 30209610
- [Derived] Tyberg A, Sharaiha RZ, Kedia P, Kumta N, Gaidhane M, Artifon E, Giovannini M, Kahaleh M. EUS-guided pancreatic drainage for pancreatic strictures after failed ERCP: a multicenter international collaborative study. Gastrointest Endosc. 2017 Jan;85(1):164-169. doi: 10.1016/j.gie.2016.07.030. Epub 2016 Jul 25. PMID 27460387
- [Derived] Kahaleh M, Perez-Miranda M, Artifon EL, Sharaiha RZ, Kedia P, Penas I, De la Serna C, Kumta NA, Marson F, Gaidhane M, Boumitri C, Parra V, Rondon Clavo CM, Giovannini M. International collaborative study on EUS-guided gallbladder drainage: Are we ready for prime time? Dig Liver Dis. 2016 Sep;48(9):1054-7. doi: 10.1016/j.dld.2016.05.021. Epub 2016 Jun 3. PMID 27328985
- [Derived] Tyberg A, Perez-Miranda M, Sanchez-Ocana R, Penas I, de la Serna C, Shah J, Binmoeller K, Gaidhane M, Grimm I, Baron T, Kahaleh M. Endoscopic ultrasound-guided gastrojejunostomy with a lumen-apposing metal stent: a multicenter, international experience. Endosc Int Open. 2016 Mar;4(3):E276-81. doi: 10.1055/s-0042-101789. PMID 27004243
- [Derived] Kedia P, Tyberg A, Kumta NA, Gaidhane M, Karia K, Sharaiha RZ, Kahaleh M. EUS-directed transgastric ERCP for Roux-en-Y gastric bypass anatomy: a minimally invasive approach. Gastrointest Endosc. 2015 Sep;82(3):560-5. doi: 10.1016/j.gie.2015.03.1913. Epub 2015 May 5. PMID 25952086